CLINICAL TRIAL: NCT04243486
Title: A Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study of the Safety and Efficacy of UHE-105 Shampoo in Subjects With Scalp Psoriasis
Brief Title: A Study of the Safety and Efficacy of UHE-105 Shampoo in Subjects With Scalp Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 188-0552-202
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Scalp Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UHE-105 Shampoo (Experimental): UHE-105 Shampoo applied topically once daily to psoriatic lesions on the scalp for up to four (4) weeks
  Interventions: Drug: UHE-105
- Vehicle Shampoo (Placebo Comparator): Vehicle Shampoo applied topically once daily to psoriatic lesions on the scalp for up to four (4) weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: UHE-105 — Topical shampoo containing active drug
  Arms: UHE-105 Shampoo
Drug: Vehicle — Topical shampoo containing no active drug
  Arms: Vehicle Shampoo

SUMMARY:
This study is to compare the safety and efficacy of UHE-105 Shampoo with that of the vehicle (VEH) Shampoo in subjects with scalp psoriasis. Half of the subjects will receive the UHE-105 Shampoo, while the other half will receive the VEH Shampoo with no active drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female 18 years of age or older.
* Subject has provided written informed consent.
* Females must be post-menopausal , surgically sterile or use an effective method of birth control. , Women of childbearing potential must have a negative urine pregnancy test at Visit 1/Baseline.
* Subject has a clinical diagnosis of stable moderate to severe scalp psoriasis affecting at least 10% of the scalp.
* Subject is willing and able to apply the test article(s) as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
* Subject, in the investigator's opinion, is in good general health and free of any disease state or physical condition that might impair evaluation of scalp psoriasis or exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject has spontaneously improving or rapidly deteriorating scalp psoriasis.
* Subject has guttate, pustular, erythrodermic, or other non-plaque forms of scalp psoriasis.
* Subject has any physical condition which, in the investigator's opinion, could impair evaluation of scalp psoriasis, adrenal axis function (e.g., Addison's Disease, Cushing's Syndrome), or which exposes the subject to an unacceptable risk by study participation.
* Subject has scalp psoriasis that necessitates systemic or other concomitant topical therapies during the study.
* Subject has a history of psoriasis unresponsive to topical treatments.
* Subject has any hair on their scalp of a length that extends beyond the subject's chin.
* Subject has any open sores, lesions, cuts, or infections, etc. on the scalp or has had a scalp surgical procedure within the past 30 days.
* Subject is currently enrolled in an investigational drug or device study.

Other protocol defined inclusion or exclusion criteria assessed by the study staff may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment (IGA) Treatment Success | Day 15
  The percentage of subjects classified as IGA treatment success
Investigator's Global Assessment (IGA) Treatment Success | Day 29
  The percentage of subjects classified as IGA treatment success

SECONDARY OUTCOMES:
Clinical signs of psoriasis (scaling, erythema and plaque elevation) Treatment Success | Days 8, 15, and 29
  Percentage of subjects classified as treatment success for each of the clinical signs of psoriasis (scaling, erythema and plaque elevation)
Change in Percentage of scalp affected by psoriasis | Days 8, 15, and 29
  Change from baseline in the percentage of scalp affected by psoriasis
Percentage of subjects with pruritus severity score treatment success | Days 8, 15, and 29
  Percentage of subjects classified as treatment success for change from baseline in pruritus severity score using an 11-point numeric rating scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Andrasfay, Study Director — Therapeutics, Inc.
Locations (2):
- United States (2):
  - 01, San Diego, California
  - 02, High Point, North Carolina

IPD SHARING:
Plan to Share IPD: No